CLINICAL TRIAL: NCT00005909
Title: Clinical, Biochemical, and Molecular Investigations Into Alkaptonuria
Brief Title: Study of Alkaptonuria
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000141; 00-HG-0141
Record Dates: First submitted 2000-06-13; First posted 2000-06-14 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-19

CONDITIONS: Alkaptonuria
Keywords: Homogentisic Acid; Ochronosis; Inborn Error of Metabolism; Arthritis; Enzyme Defect; Natural History; Alkaptonuria
MeSH Terms: conditions — Alkaptonuria; Ochronosis; Metabolism, Inborn Errors; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alkaptonuria: Patients with confirmed or suspected alkaptonuria

SUMMARY:
The purpose of this study is to gain a better understanding of alkaptonuria and collect medical data on patients who may later participate in new drug trials for this rare genetic disease. In alkaptonuria, a pigment called homogentisic acid collects in bone and connective tissue, causing arthritis and eventually bone fractures, and also causes discoloration in the ears and whites of the eyes. Some patients also develop kidney stones and heart valve problems. Alkaptonuria has not been studied for decades; and scientists expect to gain comprehensive clinical information using current medical techniques.

Patients with alkaptonuria who are at least two years of age may be eligible for this study. Participants will be evaluated at NIH s Clinical Center for 3 to 5 days every 2 to 3 years. They will have a medical history, physical examination, routine blood and urine tests. Blood may also be collected to measure a type of collagen that indicates new bone formation and to analyze DNA for genetic studies. 24-hour urine collections will be done to measure organic acids and homogentisic acid excretion, assess overall kidney function, and evaluate bone metabolism. A total of 89.5 ml (about 6 tablespoons) of blood will be drawn for these studies in adults and 51 ml (about 3 tablespoons) in children.

Patients will (may) also have bone X-rays, kidney ultrasound, brain and chest computerized tomography (CT) scans, magnetic resonance imaging (MRI) scans of affected joints, electrocardiograms, echocardiogram, lung function tests, and a hearing test. Photographs of the face and full body (with underwear on) will be taken.

As medically indicated, patients will also have consultations with dentistry and ophthalmology, with physical therapy and rehabilitation medicine for arthritis management, and with cardiology for heart valve evaluation. When appropriate, patients may also have dermatology, pulmonology and neurology consultations.

The information from this study will enable doctors to better advise patients with alkaptonuria about their disease and treatment options. It will also prepare the way for clinical studies of a new drug that blocks production of homogentisic acid.

DETAILED DESCRIPTION:
Alkaptonuria is a rare autosomal recessive disorder in which homogentisic acid accumulates and destroys connective tissue and bone, creating a condition called ochronosis. Symptoms generally begin in the third or fourth decade and progress to incapacitating spondylosis, arthropathy, and fractures by the sixth to eighth decades. Cardiac valve deterioration and renal and prostate calculi also occur. Diagnosis is made by measurement of gram quantities of urinary homogentisic acid, which turns black on alkali treatment or exposure to oxygen. In the body, homogentisic acid forms a characteristic blue color in the cartilage of the ear and brown color in the sclera of the eye. The gene for homogentisic acid oxidase was isolated in 1996, and scores of different mutations have been defined. Only symptomatic treatment is available. We propose to investigate up to 300 alkaptonuria patients, particularly adults, every 2-3 years during 3-5 day admissions, to define the disorder using current medical techniques. We will use our expertise in this disease to advise the population in terms of prognosis and therapy. Mutation analysis, with correlation of genotype and phenotype, will be performed as a secondary goal. Finally, we will work to identify suitable clinical outcome measures that may be useful for future trials. The present protocol does not include treatment with nitisinone. Instead, we will examine patients, measure baseline excretion of homogentisic acid on 24-hour urine, and characterize the signs and symptoms of alkaptonuria at different ages.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients entering this study will carry the diagnosis of alkaptonuria, although we will confirm this diagnosis during the admission. Alkaptonuria has been reported to occur throughout the world, with concentrations in the Dominican Republic, Slovakia, and Germany. We plan to recruit patients of all ethnic backgrounds.

EXCLUSION CRITERIA:

Patients will be excluded if they cannot travel to the NIH due to their medical condition or are in imminent danger of death due to, e.g., cardiac involvement. Children under two years of age are excluded because they are virtually never affected with the symptoms of this disorder, and their investigations can be delayed.

Ages: 2 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed or suspected alkaptonuria@@@
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2000-06-21 (Actual)

PRIMARY OUTCOMES:
To delineate the clinical and laboratory findings of alkaptonuria, using state-of-the-art medical technology such as cardiac CT, MRI, and echocardiograms. | Ongoing
  To delineate the clinical and laboratory findings of alkaptonuria, using state-of-the-art medical technology such as cardiac CT, MRI, and echocardiograms.

SECONDARY OUTCOMES:
To understand the natural history and rates of progression to identify suitable outcome measures for future studies. | Ongoing
  To understand the natural history and rates of progression to identify suitable outcome measures for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Introne, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This data will be deidentified.
Supporting Information: Study Protocol
Time Frame: While the study is open.
Access Criteria: All data sharing will be approved by the NHGRI Tech Transfer Office.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-HG-0141.html